CLINICAL TRIAL: NCT01458405
Title: Randomized, Double-Blind, Placebo-Controlled Phase I/II Study of the Safety and Efficacy of Intracoronary Delivery of Allogeneic Cardiosphere-Derived Cells in Patients With a Myocardial Infarction and Ischemic Left Ventricular Dysfunction
Brief Title: Allogeneic Heart Stem Cells to Achieve Myocardial Regeneration
Acronym: ALLSTAR
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: On February 28, 2019, Capricor ceased ongoing follow-up activities and terminated the ALLSTAR trial to focus resourcing on its active CAP-1002 program, HOPE-2.
Sponsor: Capricor Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002-01; RC3HL103356-01 (NIH)
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-02

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Heart Attack; Stem cell; Left ventricular dysfunction; Congestive heart failure
MeSH Terms: conditions — Myocardial Infarction; Ventricular Dysfunction, Left; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- CAP-1002 Allogeneic Cardiosphere-Derived Cells (Active Comparator)
  Interventions: Biological: CAP-1002 Allogeneic Cardiosphere-Derived Cells

INTERVENTIONS:
Biological: CAP-1002 Allogeneic Cardiosphere-Derived Cells — Single dose, blinded, intracoronary infusion of 25 Million cardiosphere-derived cells
  Arms: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Drug: Placebo — Single, blinded, intracoronary infusion of a placebo solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Allogeneic Cardiosphere-Derived Cells (CAP-1002) is safe and effective in decreasing infarct size in patients with a myocardial infarction.

ELIGIBILITY:
Inclusion Criteria

1. History of MI (STEMI or NSTEMI) within the prior 12 months due to a coronary artery event and evidenced by at least two of the following: typical ischemic symptoms, serial ST-T changes (new ST elevation or new left bundle block) and/or elevated troponin or Creatine phosphokinase MB isoenzyme (CK-MB) >5 times the upper limit of normal. Also at least one of the following: development of pathological Q wave ECG changes, imaging evidence of new loss of viable myocardium, or new regional wall motion abnormalities.
2. History of percutaneous coronary intervention (PCI), with stent placement resulting in Thrombolysis in Myocardial Infarction (TIMI) flow = 3, in the coronary artery supplying the infarcted, dysfunctional territory and through which the treatment will be infused.
3. At least one assessment of left ventricular ejection function (LVEF) <=0.45 as determined by any one of the standard modalities (echocardiography, ventriculography, nuclear imaging, CT and/or MRI) prior to or during the screening period.

   * For participants that fulfill the criteria of Recent MI (i.e., within 90 days of MI) at time of screening visit: assessment must be post-reperfusion after index MI and the most recent test prior to or during the screening period.
   * For participants that fulfill the criteria of Chronic MI (i.e., greater than 90 days from MI) at the time of screening visit: assessment must be at least 21 days post-reperfusion after index MI and the most recent test prior to or during the screening period.

   Note: participants may screen as a Recent MI but be randomized into the Chronic MI strata if the infusion date is > 90 days post-MI.
4. Left ventricular infarct size of >= 15% of left ventricular mass in the qualifying infarct-related region to be infused as determined by centrally read screening MRI, with associated thinning and/or hypokinesis, akinesis, or dyskinesis, with no large aneurysmal area in the infarcted regions.
5. No further revascularization clinically indicated at the time the participants is assessed for participation in the clinical trial.
6. Ability to provide informed consent and follow-up with protocol procedures.
7. Age >= 18 years.

Exclusion Criteria

1. Participants with a history of coronary artery bypass surgery, and a patent graft (arterial or saphenous vein graft) attached to the coronary artery to be infused.
2. Diagnosed or suspected myocarditis.
3. History of cardiac tumor, or cardiac tumor demonstrated on screening MRI.
4. History of acute coronary syndrome in the 4 weeks prior to study infusion.
5. History of previous stem cell therapy.
6. History of radiation treatment to the central or left side of thorax.
7. Current or history (within the previous 5 years) of systematic auto-immune or connective tissue disease including, but not limited to, giant cell myocarditis, cardiac or systemic sarcoidosis, Dressler's syndrome, chronic recurrent or persistent pericarditis.
8. History of or current treatment with immunosuppressive, anti-inflammatory, or other agents to treat manifestations of systemic immunologic reactions, including chronic systemic corticosteroids, biologic agents targeting the immune system, anti-tumor and anti-neoplastic drugs, anti-vascular endothelial growth factor, or chemotherapeutic agents within 3 months prior to enrollment.
9. Prior implantable cardioverter defibrillator (ICD) and/or pacemaker placement where study imaging site has not been trained and certified specifically for this protocol to conduct cardiac MRI in participants with ICD and/or pacemaker placement.

   a. Presence of a pacemaker and/or ICD generator with any of the following limitations/conditions are excluded: i. Manufactured before the year 2000, ii. Leads implanted < 6 weeks prior to signing informed consent, iii. Non-transvenous epicardial, abandoned, or no-fixation leads, iv. Subcutaneous ICDs, v. Leadless pacemakers, vi. Any other condition that, in the judgement of device-trained staff, would deem an MRI contraindicated.

   b. Pacemaker dependence with an ICD (Note: pacemaker-dependent candidates without an ICD are not excluded).

   c. A cardiac resynchronization therapy (CRT) device implanted < 3 months prior to signing informed consent.
10. Estimated glomerular filtration rate < 30 mL/min.
11. Participation in an on-going protocol studying an experimental drug or device, or participation in an interventional clinical trial within the last 30 days.
12. Diagnosis of arrhythmogenic right ventricular cardiomyopathy.
13. Current alcohol or drug abuse.
14. Pregnant/nursing women and women of child-bearing potential that do not agree to use at least two forms of active and highly reliable method(s) of contraception. Acceptable methods of contraception include contraceptive pills, depo-progesterone injections, a barrier contraceptive such as a condom with or without spermicide cream or gel, diaphragms or cervical cap with or without spermicide or gel, or an intrauterine device (IUD).
15. Human Immunodeficiency Virus (HIV) infection.
16. Viral hepatitis.
17. Uncontrolled diabetes (HbA1c>9%).
18. Abnormal liver function (Serum Glutamic Pyruvic Transaminase/Alanine aminotransferase > 3 times the upper reference range) and/or abnormal hematology (hematocrit < 25%, White Blood Cell < 3000 µl, platelets < 100,000 µl) studies without a reversible, identifiable cause.
19. Sustained ventricular tachycardia (VT) or non-sustained ventricular tachycardia > 30 beats, not associated with the acute phase of a previous MI (> 48 hours after the MI onset) or a new acute ischemic episode.
20. Ventricular fibrillation not associated with a new acute ischemic episode.
21. New York Heart Association (NYHA) Class IV congestive heart failure.
22. Evidence of tumor on screening chest/abdominal/pelvic (body) CT scan.
23. Any prior transplant.
24. Known hypersensitivity to dimethyl sulfoxide (DMSO).
25. Known hypersensitivity to bovine products.
26. Any malignancy within 5 years (except for in-situ non-melanoma skin cancer and in-situ cervical cancer) of signing the informed consent form.
27. Any condition or other reason that, in the opinion of the Investigator or Medical Monitor, would render the participants unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-11-13 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Litvack, MD, Study Director — Capricor Inc.
Locations (32):
- United States (32):
  - Cardiology, P.C., Birmingham, Alabama
  - Heart Center Research, Huntsville, Alabama
  - Scripps, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida - Shands Hospital, Gainesville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Prairie Heart - St. John's Hospital, Springfield, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Michigan CardioVascular Institute, Saginaw, Michigan
  - Metropolitan Heart and Vascular Institute / Mercy Hospital, Coon Rapids, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University at Buffalo, Buffalo, New York
  - Lenox Hill Hospital, New York, New York
  - Carolinas HealthCare System, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - SUMMA Health System, Akron, Ohio
  - Lindner Center for Research and Education at the Christ Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Austin Heart, Austin, Texas
  - University of Texas Memorial Hermann Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Swedish Medical Center - Heart and Vascular Research, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Aurora Research Institute, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Ostovaneh MR, Makkar RR, Ambale-Venkatesh B, Ascheim D, Chakravarty T, Henry TD, Kowalchuk G, Aguirre FV, Kereiakes DJ, Povsic TJ, Schatz R, Traverse JH, Pogoda J, Smith RD, Marban L, Marban E, Lima JAC. Effect of cardiosphere-derived cells on segmental myocardial function after myocardial infarction: ALLSTAR randomised clinical trial. Open Heart. 2021 Jul;8(2):e001614. doi: 10.1136/openhrt-2021-001614. PMID 34233913
- [Derived] Makkar RR, Kereiakes DJ, Aguirre F, Kowalchuk G, Chakravarty T, Malliaras K, Francis GS, Povsic TJ, Schatz R, Traverse JH, Pogoda JM, Smith RR, Marban L, Ascheim DD, Ostovaneh MR, Lima JAC, DeMaria A, Marban E, Henry TD. Intracoronary ALLogeneic heart STem cells to Achieve myocardial Regeneration (ALLSTAR): a randomized, placebo-controlled, double-blinded trial. Eur Heart J. 2020 Sep 21;41(36):3451-3458. doi: 10.1093/eurheartj/ehaa541. PMID 32749459

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants at 30 active sites between 13 November 2012 to 03 July 2017. Study had 2 phases: Phase 1 (safety cohort) and Phase 2 (randomized double-blind cohort).
Pre-assignment Details: After completion of screening procedures, and at least 4 weeks after myocardial infarction (MI), eligible Phase 1 participants received CAP-1002. In Phase 2, participants were randomized in 2:1 ratio to receive treatment with either CAP-1002 or placebo. Based on available clinical data at time of analysis, Sponsor decided not to pursue development of CAP-1002 in this indication; hence trial was stopped. Outcome measures data was planned to be collected and reported for Phase 2 part of study.
Groups:
- Phase 1: Safety Cohort:12.5 M CDCs: Participants with recent MI (defined as index MI more than 4 weeks but within 90 days prior to infusion), and chronic MI (defined as index MI more than 90 days but less than 12 months prior to infusion), randomized in safety cohort received a single infusion of CAP-1002(12.5 million [M] cells) suspended in cryopreservation solution on Day 0 and were followed up for 12 months post-infusion.
- Phase 1: Safety Cohort: 25 M CDCs: Participants with recent MI (defined as index MI more than 4 weeks but within 90 days prior to infusion), and chronic MI (defined as index MI more than 90 days but less than 12 months prior to infusion), randomized in safety cohort received a single infusion of CAP-1002 (25 M cells) suspended in cryopreservation solution on Day 0 and were followed up for 12 months post-infusion.
- Phase 2: Randomized Treatment Cohort: Placebo: Participants with recent MI (defined as index MI more than 4 weeks but within 90 days prior to infusion), and chronic MI (defined as index MI more than 90 days but less than 12 months prior to infusion), randomized to placebo received an infusion of 11.1 milliliters (mL) of cryopreservation solution on Day 0 and were followed up for 12 months post-infusion.
- Phase 2: Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells: Participants with recent MI (defined as index MI more than 4 weeks but within 90 days prior to infusion), and chronic MI (defined as index MI more than 90 days but less than 12 months prior to infusion), randomized to active treatment received a single infusion of CAP-1002 (25 M cells) suspended in cryopreservation solution on Day 0 and were followed up for 12 months post-infusion.
Period: Phase 1 (up to 12 Months)
Arm/Group | Phase 1: Safety Cohort:12.5 M CDCs | Phase 1: Safety Cohort: 25 M CDCs | Phase 2: Randomized Treatment Cohort: Placebo | Phase 2: Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Started | 4 | 10 | 0 | 0
Completed | 4 | 9 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0
Period: Phase 2 (up to 12 Months)
Arm/Group | Phase 1: Safety Cohort:12.5 M CDCs | Phase 1: Safety Cohort: 25 M CDCs | Phase 2: Randomized Treatment Cohort: Placebo | Phase 2: Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Started | 0 | 0 | 44 (Phase 1 and Phase 2 are separate populations.) | 77 (Phase 1 and Phase 2 are separate populations.)
Completed | 0 | 0 | 33 | 54
Not Completed | 0 | 0 | 11 | 23
Not completed — Study discontinued by Sponsor | 0 | 0 | 11 | 20
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population that included all participants who received investigational product.
Groups:
- Phase 1: Safety Cohort:12.5 M CDCs: Participants with recent MI (defined as index MI more than 4 weeks but within 90 days prior to infusion), and chronic MI (defined as index MI more than 90 days but less than 12 months prior to infusion), randomized in safety cohort received a single infusion of CAP-1002 (12.5 M cells) suspended in cryopreservation solution on Day 0 and were followed up for 12 months post-infusion.
- Phase 2: Randomized Treatment Cohort: Placebo: Participants with recent MI (defined as index MI more than 4 weeks but within 90 days prior to infusion), and chronic MI (defined as index MI more than 90 days but less than 12 months prior to infusion), randomized to placebo received an infusion of 11.1 mL of cryopreservation solution on Day 0 and were followed up for 12 months post-infusion.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Safety Cohort:12.5 M CDCs | Phase 1: Safety Cohort: 25 M CDCs | Phase 2: Randomized Treatment Cohort: Placebo | Phase 2: Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells | Total
Number analyzed (Participants) | 4 | 10 | 44 | 77 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 10 | 44 | 77 | 135
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 6 | 10 | 17
  Male | 4 | 9 | 38 | 67 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 7 | 7 | 15
  White | 4 | 8 | 36 | 67 | 115
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Any of the Adjudicated Events
Description: Adjudicated Events reported included: Acute myocarditis; Death due to ventricular tachycardia (VT) or ventricular fibrillation (VF); Sudden unexpected death (defined as occurring within one hour of symptom onset, or un- witnessed death); and Major adverse cardiac event (MACE) (defined as the composite incidence of death, non- fatal recurrent MI, hospitalization for heart failure, emergency room treatment for heart failure, left ventricular assist device [LVAD] placement or heart transplant).
Time Frame: Within 1-month post-infusion
Population: Analysis was performed on safety population that included all participants who received investigational product. Data this outcome measure was not planned to be collected and reported for Phase 1 part of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Treatment Cohort: Placebo: Participants with recent MI (defined as index MI more than 4 weeks but within 90 days prior to infusion), and chronic MI (defined as index MI more than 90 days but less than 12 months prior to infusion), randomized to placebo received an infusion of 11.1 mL of cryopreservation solution on Day 0 and were followed up for 12 months post-infusion.
- Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells: Participants with recent MI (defined as index MI more than 4 weeks but within 90 days prior to infusion), and chronic MI (defined as index MI more than 90 days but less than 12 months prior to infusion), randomized to active treatment received a single infusion of CAP-1002 (25 M cells) suspended in cryopreservation solution on Day 0 and were followed up for 12 months post-infusion.
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 44 | 77
Participants
  Acute myocarditis | 0 | 0
  Death due to VT/VF | 0 | 0
  Sudden unexpected death | 0 | 0
  MACE | 0 | 0

2. Primary Outcome: Percent Change From Baseline in Myocardium Mass Infarct Size at Month 12
Description: Infarct size, expressed as a percentage, was calculated by dividing the sum of infarct areas from all sections by the sum of left ventricular (LV) areas from all sections (including those without infarct scar) and multiplying by 100. Percent improvement in infarct size defined by scar as a percent of LV mass was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 12
Population: Analysis was performed on Modified Intent-to-Treat (mITT) population that included all participants in the primary randomization cohort who received investigational product, had a baseline observation, and at least one post-baseline observation. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. Data for this outcome measure was not planned to be collected and reported for Phase 1 part of the study.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 28 | 46
percent change | -7.11 (12.218) | -8.80 (10.645)
Statistical Analysis 1: Comparison: Randomized Treatment Cohort: Placebo vs Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells; Test type: Superiority; p = 0.6453, Regression, Linear — Repeated measures multivariable linear regression with Baseline as a covariate and unstructured covariance

3. Secondary Outcome: Number of Participants Experiencing Any of the Adjudicated Events
Description: Adjudicated Events reported included: Acute myocarditis; Death due to VT or VF; Sudden unexpected death (defined as occurring within one hour of symptom onset, or un- witnessed death); MACE (defined as the composite incidence of death, non- fatal recurrent MI, hospitalization for heart failure, emergency room treatment for heart failure, LVAD placement or heart transplant); New cardiac tumor formation on MRI imaging; Any hospitalization due to cardiovascular cause; Any inter-current cardiovascular illness or one related to CAP-1002 or placebo infusion, which prolongs hospitalization; New thrombolysis in myocardial infarction (TIMI) flow <=1; Development of, or an increase in frequency of VT; Development of increased anti-human leukocyte antigen (anti-HLA) antibody levels (mean fluorescence intensity [MFI] >= 1000; 5000) with development of sensitization to HLA antigens specific to CAP-1002 cardiosphere-derived cells donor.
Time Frame: Up to Month 12 post-infusion
Population: Analysis was performed on safety population that included all participants in the primary randomization cohort who received investigational product. Data for this outcome measure was not planned to be collected and reported for Phase 1 part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 44 | 77
Participants
  Acute myocarditis | 0 | 0
  Death due to VT/VF | 0 | 0
  Sudden unexpected death | 0 | 0
  MACE | 5 | 5
  Cardiac tumor | 0 | 0
  CV hospitalization | 7 | 10
  Prolonged CV hospitalization | 0 | 0
  TIMI <= 1 | 0 | 0
  VT | 1 | 0
  Donor-specific antibody, MFI >= 1000 | 3 | 5
  Donor-specific antibody, MFI >= 5000 | 1 | 1

4. Secondary Outcome: Absolute Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Month 6 and 12
Description: LVEF is the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume). LVEF expressed as percentage ejection fraction was assessed by magnetic resonance imaging. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and reported for Phase 1 part of the study.
Measure: Mean (Standard Deviation); unit: percent change ejection fraction
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
percent change ejection fraction
  Month 6: number analyzed (Participants) | 41 | 71
  Month 6 | 0.17 (3.484) | -0.02 (4.435)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | 0.01 (4.089) | -0.62 (5.239)

5. Secondary Outcome: Percent Change From Baseline in Left Ventricular Ejection Fraction (LVEF) at Month 6 and 12
Description: LVEF is the fraction of chamber volume ejected in systole (stroke volume) in relation to the volume of the blood in the ventricle at the end of diastole (end-diastolic volume). Percent change in LVEF was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
percent change
  Month 6: number analyzed (Participants) | 41 | 71
  Month 6 | 0.82 (10.890) | 0.61 (11.894)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | 0.01 (10.228) | -1.04 (13.956)

6. Secondary Outcome: Absolute Change From Baseline in Left Ventricular End Diastolic Volume (LVEDV) at Month 6 and 12
Description: LVEDV is the amount of blood in the heart's left ventricle just before the heart contracts. LVEDV was assessed by magnetic resonance imaging. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
milliliters (mL)
  Month 6: number analyzed (Participants) | 41 | 71
  Month 6 | 11.75 (23.129) | 3.92 (23.692)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | 7.59 (27.551) | 4.04 (30.511)

7. Secondary Outcome: Percent Change From Baseline in Left Ventricular End Diastolic Volume (LVEDV) at Month 6 and 12
Description: LVEDV is the amount of blood in the heart's left ventricle just before the heart contracts. Percent change in LVEDV was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
percent change
  Month 6: number analyzed (Participants) | 41 | 71
  Month 6 | 5.64 (10.742) | 2.02 (11.203)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | 4.68 (12.910) | 2.54 (13.831)

8. Secondary Outcome: Absolute Change From Baseline in Left Ventricular End Systolic Volume (LVESV) at Month 6 and 12
Description: LVESV is the amount of blood remaining in the ventricle at the end of systole, after the heart has contracted. LVESV was assessed by magnetic resonance imaging. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
mL
  Month 6: number analyzed (Participants) | 41 | 71
  Month 6 | 6.96 (17.390) | 2.63 (19.000)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | 4.51 (21.213) | 3.89 (25.476)

9. Secondary Outcome: Percent Change From Baseline in Left Ventricular End Systolic Volume (LVESV) at Month 6 and 12
Description: LVESV is the amount of blood remaining in the ventricle at the end of systole, after the heart has contracted. Percent change in LVESV was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
percent change
  Month 6: number analyzed (Participants) | 41 | 71
  Month 6 | 5.41 (11.928) | 2.34 (14.257)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | 4.77 (15.764) | 4.13 (18.572)

10. Secondary Outcome: Percent Change From Baseline in Myocardium Mass Infarct Size at Month 6 and 12
Description: Infarct size, expressed as a percentage, was calculated by dividing the sum of infarct areas from all sections by the sum of LV areas from all sections (including those without infarct scar) and multiplying by 100. Improvement in infarct size as a percent of LV mass was assessed by magnetic resonance imaging.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
percent change
  Month 6: number analyzed (Participants) | 41 | 70
  Month 6 | -0.81 (2.109) | -1.05 (1.699)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | -1.31 (2.684) | -1.83 (2.432)

11. Secondary Outcome: Absolute Change From Baseline in Infarct Size (Scar Tissue Mass) at Month 6 and 12
Description: Infarct size in grams was assessed by magnetic resonance imaging. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
grams
  Month 6: number analyzed (Participants) | 41 | 70
  Month 6 | -1.72 (2.831) | -1.66 (2.927)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | -2.57 (4.858) | -2.87 (4.256)

12. Secondary Outcome: Percent Change From Baseline in Infarct Size (Scar Tissue Mass) at Month 6 and 12
Description: Percent change in infarct size was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
percent change
  Month 6: number analyzed (Participants) | 41 | 70
  Month 6 | -5.14 (8.481) | -4.67 (7.826)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | -8.50 (13.191) | -8.86 (11.249)

13. Secondary Outcome: Absolute Change From Baseline in Viable Mass at Month 6 and 12
Description: Viable mass expressed in grams was assessed by magnetic resonance imaging. Myocardial viable mass refers to myocardial cells that are alive after myocardial injury, according to cellular, metabolic and contractile functions. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
grams
  Month 6: number analyzed (Participants) | 41 | 70
  Month 6 | 2.40 (9.780) | 0.95 (8.143)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | 1.48 (11.800) | 0.96 (9.063)

14. Secondary Outcome: Percent Change From Baseline in Viable Mass at Month 6 and12
Description: Percent change in viable mass was assessed by magnetic resonance imaging. Myocardial viable mass refers to myocardial cells that are alive after myocardial injury, according to cellular, metabolic and contractile functions. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
percent change
  Month 6: number analyzed (Participants) | 41 | 70
  Month 6 | 2.54 (10.804) | 1.07 (7.698)
  Month 12: number analyzed (Participants) | 28 | 46
  Month 12 | 2.79 (10.635) | 1.31 (7.795)

15. Secondary Outcome: Absolute Change From Baseline in Function of the Region Receiving CAP-1002 Therapy at Month 6 and 12
Description: The regions assessed of the heart were: Anterior, Lateral, Inferior and Septal. Tissue mass recovery in the function of region receiving therapy expressed as percentage improvement was assessed by magnetic resonance imaging. Absolute change was calculated as: post-baseline value-Baseline value.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
percent change
  Anterior: Month 6: number analyzed (Participants) | 41 | 70
  Anterior: Month 6 | 1.21 (8.562) | -0.61 (7.260)
  Anterior: Month 12: number analyzed (Participants) | 28 | 44
  Anterior: Month 12 | 0.53 (6.966) | -1.90 (8.681)
  Lateral: Month 6: number analyzed (Participants) | 41 | 70
  Lateral: Month 6 | -0.21 (4.731) | -0.03 (3.857)
  Lateral: Month 12: number analyzed (Participants) | 28 | 44
  Lateral: Month 12 | -0.98 (4.510) | -1.15 (3.727)
  Inferior: Month 6: number analyzed (Participants) | 41 | 70
  Inferior: Month 6 | 0.39 (5.707) | -0.68 (4.736)
  Inferior: Month 12: number analyzed (Participants) | 28 | 44
  Inferior: Month 12 | -0.78 (6.255) | -0.53 (5.614)
  Septal: Month 6: number analyzed (Participants) | 41 | 70
  Septal: Month 6 | -1.51 (5.275) | -1.52 (4.851)
  Septal: Month 12: number analyzed (Participants) | 28 | 44
  Septal: Month 12 | -2.48 (4.948) | -1.97 (6.445)

16. Secondary Outcome: Percent Change From Baseline in Function of the Region Receiving CAP-1002 Therapy at Month 6 and 12
Description: The regions assessed of the heart were: Anterior, Lateral, Inferior and Septal. Tissue mass recovery in the function of region receiving therapy expressed as percentage improvement was assessed by magnetic resonance imaging. Percent change from Baseline was calculated as: Percent change = (post-baseline value-Baseline value)/Baseline value *100%.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 42 | 74
percent change
  Anterior: Month 6: number analyzed (Participants) | 41 | 70
  Anterior: Month 6 | 6.50 (33.009) | 2.99 (42.147)
  Anterior: Month 12: number analyzed (Participants) | 28 | 44
  Anterior: Month 12 | 2.33 (18.196) | -0.39 (42.897)
  Lateral: Month 6: number analyzed (Participants) | 41 | 70
  Lateral: Month 6 | 15.18 (79.223) | 15.09 (61.698)
  Lateral: Month 12: number analyzed (Participants) | 28 | 44
  Lateral: Month 12 | 178.68 (940.725) | 15.29 (91.948)
  Inferior: Month 6: number analyzed (Participants) | 41 | 69
  Inferior: Month 6 | 14.74 (64.941) | 14.61 (86.589)
  Inferior: Month 12: number analyzed (Participants) | 28 | 43
  Inferior: Month 12 | 23.83 (131.511) | 78.79 (382.480)
  Septal: Month 6: number analyzed (Participants) | 41 | 70
  Septal: Month 6 | -3.17 (15.117) | 1.41 (42.721)
  Septal: Month 12: number analyzed (Participants) | 28 | 44
  Septal: Month 12 | -7.77 (14.477) | 6.22 (75.838)

17. Secondary Outcome: Change From Baseline in Six-Minute Walk Test at Month 6 and 12
Description: The six-minute walk test measures the distance a participant is able to walk over a total of six minutes on a hard, flat surface. The goal is for the participant to walk as far as possible in six minutes. The participant is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. The total distance walked, in meters, was recorded for each participant. Longer distances indicate better outcomes.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 43 | 77
meters
  Month 6: number analyzed (Participants) | 42 | 77
  Month 6 | 40.7 (92.49) | 15.5 (108.43)
  Month 12: number analyzed (Participants) | 32 | 53
  Month 12 | 10.5 (91.45) | 25.4 (90.08)

18. Secondary Outcome: Change From Baseline in Minnesota Living With Heart Failure Questionnaire (MLHFQ) Total Score at Month 6 and 12
Description: Health related quality of life is measured using the Minnesota Living with Heart Failure questionnaire (MLHFQ). The MLHFQ is a patient-reported outcome to measure the patient's perceptions of the influence of heart failure on physical and emotional aspects of life. The questionnaire has 21 items to assess the impact of frequent physical symptoms of heart failure and the effects of heart failure on physical and emotional functions. Responses are recorded on six-point Likert scales, ranging from 0 (none) to 5 (very much). Total Scores are summed to a range of 0-105, in which with higher scores indicate worse health-related quality of life.
Time Frame: Baseline, Month 6 and Month 12
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and reported for Phase 1 part of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 44 | 77
score on a scale
  Month 6 | -5.27 (18.195) | -8.30 (15.951)
  Month 12: number analyzed (Participants) | 32 | 53
  Month 12 | -8.47 (16.580) | -8.89 (20.636)

19. Secondary Outcome: Change From Baseline in Short Form (36) (SF-36) Scale Score at Month 6 and 12
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of participant health. The SF-36 consists of eight scaled scores (Physical Function, Physical Health, Emotional Problems, Energy/Fatigue, Emotional Well-Being, Social Functioning, Pain Scale and General Health) which are the weighted sums of the questions in their section. Each component on the SF-36 Item Health Survey is scored from 0-100 with higher scores reflecting better participant status.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 44 | 77
score on a scale
  Physical Function Scale: Month 6 | 7.84 (19.392) | 6.79 (17.041)
  Physical Function Scale: Month 12: number analyzed (Participants) | 32 | 53
  Physical Function Scale: Month 12 | 3.91 (13.182) | 6.16 (19.943)
  Physical Health Scale: Month 6 | 15.72 (34.393) | 26.08 (46.680)
  Physical Health Scale: Month 12: number analyzed (Participants) | 32 | 53
  Physical Health Scale: Month 12 | 21.09 (38.683) | 37.42 (41.171)
  Emotional Problems Scale: Month 6 | 3.03 (31.185) | 8.23 (41.237)
  Emotional Problems Scale: Month 12: number analyzed (Participants) | 32 | 53
  Emotional Problems Scale: Month 12 | 11.46 (41.139) | 12.58 (32.176)
  Energy/Fatigue Scale: Month 6 | 4.55 (20.877) | 7.29 (18.984)
  Energy/Fatigue Scale: Month 12: number analyzed (Participants) | 32 | 53
  Energy/Fatigue Scale: Month 12 | 8.59 (23.044) | 8.87 (20.254)
  Emotional Well-Being Scale: Month 6 | 2.55 (14.794) | 2.18 (14.833)
  Emotional Well-Being Scale: Month 12: number analyzed (Participants) | 32 | 53
  Emotional Well-Being Scale: Month 12 | 0.50 (17.996) | 0.72 (13.074)
  Social Functioning Scale: Month 6 | 8.24 (20.163) | 5.68 (24.379)
  Social Functioning Scale: Month 12: number analyzed (Participants) | 32 | 53
  Social Functioning Scale: Month 12 | 8.59 (18.632) | 9.91 (27.228)
  Pain Scale: Month 6 | 0.68 (22.022) | -1.01 (21.773)
  Pain Scale: Month 12: number analyzed (Participants) | 32 | 53
  Pain Scale: Month 12 | 2.50 (21.166) | 1.04 (21.447)
  General Health Scale: Month 6 | 1.36 (15.971) | 0.19 (17.100)
  General Health Scale: Month 12: number analyzed (Participants) | 32 | 53
  General Health Scale: Month 12 | -0.94 (16.335) | 2.74 (14.954)

20. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) Score at Month 6 and 12
Description: WPAI:SHP is a self-administered questionnaire that measures the effect of general health and symptom severity on work productivity and regular activities during the last 7 days. Four scores are derived as percent: Absenteeism, Presenteeism, Work Productivity Loss, Activity Impairment. Each of 4 scores expressed as impairment percentages with a total possible score range of 0 to 100, high percentage= more impairment, less productivity.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage impairment
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 43 | 77
percentage impairment
  Absenteeism: Month 6: number analyzed (Participants) | 26 | 45
  Absenteeism: Month 6 | -9.19 (22.910) | -4.53 (20.707)
  Absenteeism: Month 12: number analyzed (Participants) | 17 | 31
  Absenteeism: Month 12 | -11.94 (30.569) | -8.00 (22.943)
  Presenteeism: Month 6: number analyzed (Participants) | 25 | 46
  Presenteeism: Month 6 | -4.40 (22.376) | -8.48 (28.903)
  Presenteeism: Month 12: number analyzed (Participants) | 16 | 32
  Presenteeism: Month 12 | -8.75 (22.472) | -15.94 (33.201)
  Work Productivity Loss: Month 6: number analyzed (Participants) | 24 | 43
  Work Productivity Loss: Month 6 | -9.67 (25.096) | -10.21 (33.012)
  Work Productivity Loss: Month 12: number analyzed (Participants) | 15 | 30
  Work Productivity Loss: Month 12 | -14.87 (30.538) | -18.77 (36.380)
  Activity Impairment: Month 6: number analyzed (Participants) | 42 | 76
  Activity Impairment: Month 6 | -6.19 (27.670) | -10.26 (29.843)
  Activity Impairment: Month 12: number analyzed (Participants) | 31 | 53
  Activity Impairment: Month 12 | -5.81 (24.870) | -12.64 (28.090)

21. Secondary Outcome: Number of Participants With Change From Baseline in Patient Global Assessment (PGA) Score at Month 6 and 12
Description: PGA will ask participants to assess how their overall status has changed since prior to receiving the therapy. Possible PGA responses are "0=none", "1=mild", "2=moderate", "and 3=severe". Change from Baseline was calculated as lowest PGA score on scheduled visits minus PGA score at Baseline which resulted in possible ranges from -3 to +3. Decreasing scores indicate improvement.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 44 | 77
Participants
  Month 6: - 3 | 0 | 0
  Month 6: - 2 | 2 | 6
  Month 6: - 1 | 21 | 23
  Month 6: + 0 | 18 | 39
  Month 6: + 1 | 3 | 7
  Month 6: + 2 | 0 | 2
  Month 6: + 3 | 0 | 0
  Month 12: - 3: number analyzed (Participants) | 32 | 53
  Month 12: - 3 | 0 | 1
  Month 12: - 2: number analyzed (Participants) | 32 | 53
  Month 12: - 2 | 0 | 5
  Month 12: - 1: number analyzed (Participants) | 32 | 53
  Month 12: - 1 | 15 | 22
  Month 12: + 0: number analyzed (Participants) | 32 | 53
  Month 12: + 0 | 16 | 20
  Month 12: + 1: number analyzed (Participants) | 32 | 53
  Month 12: + 1 | 1 | 3
  Month 12: + 2: number analyzed (Participants) | 32 | 53
  Month 12: + 2 | 0 | 2
  Month 12: + 3: number analyzed (Participants) | 32 | 53
  Month 12: + 3 | 0 | 0

22. Secondary Outcome: Number of Participants With Change From Baseline in New York Heart Association (NYHA) Class at Month 6 and 12
Description: New York Heart Association (NYHA) Classification: Class I Subject with cardiac disease but without resulting limitations of physical activity. Class II Subjects with cardiac disease resulting in slight limitation of physical activity. Class III Subjects with cardiac disease resulting in marked limitation of physical activity. Class IV Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort. Change from Baseline was calculated as lowest NYHA score on scheduled visits minus NYHA score at Baseline which resulted in possible ranges from -3 to +3. Decreasing scores indicate improvement.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 44 | 77
Participants
  Month 6: - 3 | 1 | 0
  Month 6: - 2 | 0 | 3
  Month 6: - 1 | 13 | 24
  Month 6: 0 | 26 | 45
  Month 6: + 1 | 3 | 5
  Month 6: + 2 | 1 | 0
  Month 6: + 3 | 0 | 0
  Month 12: - 3: number analyzed (Participants) | 32 | 53
  Month 12: - 3 | 0 | 0
  Month 12: - 2: number analyzed (Participants) | 32 | 53
  Month 12: - 2 | 3 | 4
  Month 12: - 1: number analyzed (Participants) | 32 | 53
  Month 12: - 1 | 15 | 17
  Month 12: 0: number analyzed (Participants) | 32 | 53
  Month 12: 0 | 11 | 28
  Month 12: + 1: number analyzed (Participants) | 32 | 53
  Month 12: + 1 | 2 | 4
  Month 12: + 2: number analyzed (Participants) | 32 | 53
  Month 12: + 2 | 1 | 0
  Month 12: + 3: number analyzed (Participants) | 32 | 53
  Month 12: + 3 | 0 | 0

23. Secondary Outcome: Change From Baseline in N-terminal Pro-hormone Brain Natriuretic Peptide (NT-proBNP) Biomarker at Month 6 and 12
Description: NT-proBNP was the cardiac biomarkers assessed through serum sample.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 43 | 75
pg/mL
  Month 6: number analyzed (Participants) | 43 | 74
  Month 6 | -126.4 (621.45) | -361.6 (626.56)
  Month 12: number analyzed (Participants) | 31 | 50
  Month 12 | -283.2 (571.86) | -395.8 (752.83)

24. Secondary Outcome: Change From Baseline in Log Transformed N-terminal Pro-hormone Brain Natriuretic Peptide (NT-proBNP) Biomarker at Month 6 and 12
Description: NT-proBNP was the cardiac biomarkers assessed through serum sample.
Time Frame: Baseline, Month 6 and Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: log pg/mL
Arm/Group | Randomized Treatment Cohort: Placebo | Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
Number analyzed (Participants) | 43 | 75
log pg/mL
  Month 6: number analyzed (Participants) | 43 | 74
  Month 6 | -0.26 (0.732) | -0.50 (0.557)
  Month 12: number analyzed (Participants) | 31 | 50
  Month 12 | -0.46 (0.761) | -0.63 (0.616)

ADVERSE EVENTS:
Time Frame: Phase 1 and 2: Adverse Events data was collected from first infusion up to 12 Month post-infusion in each Phase of the study (i.e., up to Month 12)
Description: Analysis was performed on safety population.
Arm/Group | Phase 1: Safety Cohort:12.5 M CDCs | Phase 1: Safety Cohort: 25 M CDCs | Phase 2: Randomized Treatment Cohort: Placebo | Phase 2: Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/10 | 0/44 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/10 | 15/44 | 20/77
Other Adverse Events (participants affected / at risk) | 4/4 | 10/10 | 24/44 | 42/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Safety Cohort:12.5 M CDCs (N=4) | Phase 1: Safety Cohort: 25 M CDCs (N=10) | Phase 2: Randomized Treatment Cohort: Placebo (N=44) | Phase 2: Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells (N=77)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Angina Pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erosive Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatitis Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angiogram (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Implantable Defibrillator Insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Implantable Icd Insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intermittent Claudication (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Safety Cohort:12.5 M CDCs (N=4) | Phase 1: Safety Cohort: 25 M CDCs (N=10) | Phase 2: Randomized Treatment Cohort: Placebo (N=44) | Phase 2: Randomized Treatment Cohort: CAP-1002 Allogeneic Cardiosphere-Derived Cells (N=77)
Cardiac Failure (Cardiac disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (2) | 1 (1) | 4 (4)
Catheter Site Related Reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 6 (6) | 5 (5)
Drug Intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 2 (2) | 2 (5) | 1 (1)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant Site Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Brain Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign Body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin I Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (6) | 4 (4)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 6 (6) | 5 (5)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 3 (5) | 3 (3)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 4 (5)
Dizziness Postural (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (4) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (5) | 6 (6)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 5 (5) | 5 (5)
Anaemia Macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anginal Equivalent (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Atrial Thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular Block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular Block First Degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia And Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bundle Branch Block Left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Aneurysm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Cardiac Ventricular Thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Coronary Artery Dissection (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary Artery Thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracardiac Thrombus (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mixed Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyphaema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Catheter Site Bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic Lesion (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash Pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Tinea Pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vascular Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Implantable Defibrillator Insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous Fistula (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermittent Claudication (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ALT Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AST Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood Potassium Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Uric Acid Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ECG PR Prolongation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ECG ST Segment Depression (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ECG ST Segment Elevation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ejection Fraction Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematocrit Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver Function Test Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mean Cell Haemoglobin Conc Dec (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mean Cell Haemoglobin Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red Blood Cells Urine (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red Cell Distribution Width Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid Retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dupuytrens Contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensory Disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Libido Decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Based on available clinical data at time of the analysis, the Sponsor decided not to pursue development of CAP-1002 in this indication; hence the trial was stopped.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT01458405/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT01458405/SAP_001.pdf